CLINICAL TRIAL: NCT04683289
Title: Surgical Outcomes of Visco-Circumferential-Suture-Trabeculotomy in Primary Congenital Glaucoma: A 3-year Randomized Controlled Study
Brief Title: Visco-Circumferential-Suture-Trabeculotomy Versus Trabeculotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Visco-Suture-Trabeculotomy
Record Dates: First submitted 2020-12-19; First posted 2020-12-24 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Primary Congenital Glaucoma
MeSH Terms: conditions — Hydrophthalmos | interventions — Trabeculectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Visco-Circumferential-Suture-Trabeculotomy (Experimental): Visco-Circumferential-Suture-Trabeculotomy
  Interventions: Procedure: trabeculotomy
- viscotrabeculotomy (Active Comparator): Viscotrabeculotomy
  Interventions: Procedure: trabeculotomy

INTERVENTIONS:
Procedure: trabeculotomy — performing partial unroofing of the SC and viscoelastic injection into the 2 ostia of the canal. This was followed by connecting the scalemm canal to the anterior chamber

SUMMARY:
comparing outcomes of Visco-Circumferential-Suture-Trabeculotomy in primary congenital glaucoma to trabeculotomy

DETAILED DESCRIPTION:
prospective randomized interventional study conducted on infants below the age of 2 years with PCG attending the outpatient clinic of Mansoura Ophthalmic Center of Mansoura University were recruited to compare the long-term surgical outcomes of this proposed technique (VCST) and rigid probe VT in patients with PCG.

ELIGIBILITY:
Inclusion Criteria:

* infants below the age of 2 years with PCG

Exclusion Criteria:

* patients older than 2 years on presentation
* eyes with previous surgery
* eyes with secondary glaucoma
* eyes diagnosed as anterior segment dysgenesis syndrome

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
IOP | 36 months
  intraocular pressure measuring

SECONDARY OUTCOMES:
complications | 36 months months
  visual devastating complications

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmic Center, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No